CLINICAL TRIAL: NCT07318233
Title: Adaptive Self-Efficacy-Based AI Coaching for Enhanced Indoor Cycling Performance: A Personalized Machine Learning Approach
Brief Title: Adaptive Self-Efficacy-Based AI Coaching for Cycling
Acronym: AI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Anna Queiroz, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 20251354
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Exercise Training; Exercise Behavior; Exercise Adherence Challenges; Motivation for Physical Activity; Motivational Enhancement
Keywords: Physical Activity; AI affirmations; just-in-time adaptive intervention; cycling
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): No affirmations delivered. Participants receive only time notifications at 5, 10, 15, and 19 minutes for pacing awareness. Same equipment worn to control for potential monitoring effects.
- Group 1: Self-efficacy-based AI coaching (Experimental): The Thompson Sampling contextual bandit algorithm, trained on Session 1 data, monitors performance continuously and evaluates every 5 seconds whether to deliver an affirmation.
  Interventions: Behavioral: Group 1: Self-efficacy-based AI coaching
- Group 2: Static AI Affirmations (Active Comparator): Generic motivational messages delivered at fixed intervals (minutes 3, 6, 9, 12, 15, and 18) regardless of performance state. Messages follow the same complexity gradient based on elapsed time rather than individual response.
  Interventions: Behavioral: Group 2: Static AI Affirmations

INTERVENTIONS:
Behavioral: Group 1: Self-efficacy-based AI coaching — The Thompson Sampling contextual bandit algorithm, trained on Session 1 data, monitors performance continuously and evaluates every 5 seconds whether to deliver an affirmation. The policy is trained to maximize a multi-objective "efficacy-preserving performance" function that rewards:
  * Maintaining target power relative to rolling 30s/2min/5min baselines
  * Stabilizing short-horizon power variability (30s coefficient of variation)
  * Stabilizing heart-rate (HR) trajectory consistent with efficient pacing
  The decision process considers:
  * Current power relative to 30-second, 2-minute, and 5-minute rolling averages
  * Power output variability (coefficient of variation over past 30 seconds)
  * Heart rate trajectory and cardiac drift patterns
  * Cadence stability and changes from baseline
  * Time elapsed and expected fatigue progression based on power-duration curve Self-efficacy-based AI coaching adapts to physiological measures (power and heart rate).
  Arms: Group 1: Self-efficacy-based AI coaching
Behavioral: Group 2: Static AI Affirmations — Generic motivational messages delivered at fixed intervals (minutes 3, 6, 9, 12, 15, and 18) regardless of performance state. Messages follow the same complexity gradient based on elapsed time rather than individual response:
  * Minutes 3, 6: "You're building momentum with every pedal stroke-maintain this strong rhythm"
  * Minutes 9, 12: "Strong effort-push through this challenge"
  * Minutes 15, 18: "Final push-finish strong"
  Arms: Group 2: Static AI Affirmations

SUMMARY:
The primary objective of this study is to evaluate whether adaptive, AI-delivered personalized self-efficacy-based AI coaching based on real-time physiological and performance feedback enhance indoor cycling power output during a 20-minute time trial compared to static affirmations and exercise-only control conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years

  * Recreationally active
  * Familiar with stationary cycling
  * Able to complete 20 minutes of vigorous cycling

Exclusion Criteria:

* Cardiovascular, metabolic, or respiratory conditions

  * Medications affecting heart rate response
  * Lower extremity injury within past 3 months
  * Competitive cyclists (>10 hours cycling/week)
  * Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-23 (Estimated); Study Completion 2028-12-28 (Estimated)

PRIMARY OUTCOMES:
Mean cycling power output during 20-minute time trial | During the 20-minute time trial (collected continuously; analyzed as mean over 0-20 minutes)
  Average cycling power output over the full 20-minute time trial. The outcome compares mean power between intervention arms (adaptive AI coaching vs. static affirmations vs. exercise-only control). Power is captured continuously via the cycling ergometer and summarized as the mean watts for each participant's trial.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Queiroz, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No